CLINICAL TRIAL: NCT04102761
Title: Platelet Rich Plasma and Bone Marrow Aspirate for Lumbar Intradiscal Injections: A Multicenter Prospective Randomized Controlled Trial in Patients With Internal Disc Disruption
Brief Title: The Use of PRP and BMC in Patients With Internal Disc Disruption Multicenter Prospective Randomized Controlled Trial in Patients With Internal Disc Disruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Annu Navani (Other)
Collaborators: Andrews Research & Education Foundation (Other)
Responsible Party: Sponsor-Investigator, Annu Navani, Principal Investigator, Comprehensive Spine & Sports Center, Campbell, CA
Organization: Comprehensive Spine & Sports Center, Campbell, CA (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N003R113
Record Dates: First submitted 2018-04-17; First posted 2019-09-25 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Internal Disc Disruption

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one of three arms of the study. The first group will receive a trigger point injection of saline into the deep tissue. The second group will receive an injection of approximately 1-2 mL of Platelet RP into the painful disc/discs. The third group will receive an injection of approximately 1-2 mL of Bone Marrow Concentrate into the painful disc/discs. No more than three discs will be injected.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trigger Point Needling (Placebo Comparator): The first group will receive a deep trigger point injection of saline into deep tissue.
  Interventions: Procedure: Intradiscal PRP & BMC Injections
- Platelet Rich Plasma Injection (Active Comparator): The Platelet Rich Plasma group will receive an injection of approximately 1-2 mL of Platelet Rich Plasma into the painful disc/discs.
  Interventions: Procedure: Intradiscal PRP & BMC Injections
- Bone Marrow Aspirate Injection (Active Comparator): The third group will receive an injection of approximately 1-2 mL of Bone Marrow Concentrate into the painful disc/discs.
  Interventions: Procedure: Intradiscal PRP & BMC Injections

INTERVENTIONS:
Procedure: Intradiscal PRP & BMC Injections — The intervention to be studied is the intradiscal delivery of autologous Platelet Rich Plasma (PRP) or bone marrow concentrate (BMC) into the nucleus pulposus of the disrupted disc(s).

SUMMARY:
The condition being studied is chronic low back or leg pain in patients with internal disc disruption (IDD). The intervention to be studied is the intradiscal delivery of autologous Platelet Rich Plasma (PRP) or bone marrow concentrate (BMC) into the nucleus pulposus of the disrupted disc(s).

DETAILED DESCRIPTION:
This multi-center randomized controlled pilot trial will be the first to evaluate the response of PRP and BMC for discogenic pain by direct comparison. The investigators propose to incorporate a crossover design that compares placebo to two treatment modalities (i.e. Neutrophil-Poor PRP [NP-PRP] and BMC).

If the investigators can demonstrate statistically significant and clinically meaningful improvements in study's primary and secondary outcome measures, this study will have identified a natural, effective and sustainable treatment for discogenic back pain that currently accounts for the highest level of disability in US. This will help guide physicians in the choice of care between surgical and conservative treatment options when treating patients.

ELIGIBILITY:
Inclusion Criteria:

* A high index of suspicion for discogenic pain, i.e. painful degenerative discs with or without contained protrusions
* Age greater than 18 and less than 70 years
* Maintained intervertebral disc heights of at least 50%
* Pain not generated from facet joints, sacro-iliac joints or any pathology other than discogenic origin.
* Pain is not responsive to conservative treatment measures (oral medications, epidural steroid injections, physical therapy)
* Pain persists for an extended period of time (i.e., at least 3 months)
* High intensity zone (HIZ) in annular fissure detected on T2 or STIR MRI, degenerated discs or contained disc protrusions.
* No evidence of contraindications to undergo procedure such as pregnancy, active infection, bleeding disorder, or metastatic cancer
* English speaking

Exclusion Criteria:

* Disc extrusions, disc sequestrations, severe spinal stenosis, or severe disc degeneration with grade 5 Pfirmann index or with Modic 3 level change.
* Patient refusal
* Presence of a known bleeding disorder
* Pregnancy
* Systemic or local infection
* Presence of an unstable medical or psychiatric condition
* Prior intradiscal procedure (ie. IDET, Nucleoplasty)
* Inaccessibility to discs such as fusion
* Non-English speaking
* Prior fusion surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Worsening of Disc Pathology with Injection of Biologics | 24 weeks post procedure
  Pre and post op discs will be examined and compared for worsening pathology.
Improvement in Disc Pain with Injection of Biologics | 24 weeks post procedure
  Pre and post op Pain will be measured and compared by Numeric Rating Scale (NRS) Numeric Pain Rating Scale (NRS): Measured from 0-10, 0 minimum score (better outcome) and 10 maximum score (worse outcome) Oswestry Low back disability (ODS): Measured from 0-50, 0 minimum score and 10 maximum score. The numbers are then calculated into percentages between 0% (minimum disability- better outcome)-100% (maximum disability- worse outcome) NASS Patient satisfaction Index (NASS): Measured from 0-4, 0 (better outcome) and 4 (worse outcome)
Improvement in Function in Patients with Injection of Biologics | 24 weeks post procedure
  Pre and post op function will be measured and compared by Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Patient Satisfaction | Pre injection, 1 month post op, 3 months post op, 6 months post op, 1 year.
  Patient satisfaction will be measured by the modified North American Spine Surgery (NASS) Outcome Questionnaire
Hospitalization | Pre injection, 1 month post op, 3 months post op, 6 months post op, 1 year.
  Hospitalization will be measured by patient's self report.
Spine Surgery | Pre injection, 1 month post op, 3 months post op, 6 months post op, 1 year.
  Spine Surgery will be measured by patient's self report.
Medications | Pre injection, 1 month post op, 3 months post op, 6 months post op, 1 year.
  Medications will be measured by patient's self report.

CONTACTS AND LOCATIONS:
Overall Officials: Annu Navani, MD, Principal Investigator — Comprehensive Spine & Sports Center
Locations (4):
- United States (4):
  - Alex Hames, Campbell, California
  - The Orthohealing Center, Los Angeles, California
  - Texas Spine and Joint Hospital, Tyler, Texas
  - Nexus Pain Care, Provo, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehra M, Hill K, Nicholl D, Schadrack J. The burden of chronic low back pain with and without a neuropathic component: a healthcare resource use and cost analysis. J Med Econ. 2012;15(2):245-52. doi: 10.3111/13696998.2011.642090. Epub 2011 Dec 5. PMID 22136441
- [Background] Zhang YG, Guo TM, Guo X, Wu SX. Clinical diagnosis for discogenic low back pain. Int J Biol Sci. 2009 Oct 13;5(7):647-58. doi: 10.7150/ijbs.5.647. PMID 19847321
- [Background] Omlor GW, Nerlich AG, Tirlapur UK, Urban JP, Guehring T. Loss of notochordal cell phenotype in 3D-cell cultures: implications for disc physiology and disc repair. Arch Orthop Trauma Surg. 2014 Dec;134(12):1673-81. doi: 10.1007/s00402-014-2097-2. Epub 2014 Oct 28. PMID 25348151
- [Background] Konttinen YT, Kemppinen P, Li TF, Waris E, Pihlajamaki H, Sorsa T, Takagi M, Santavirta S, Schultz GS, Humphreys-Beher MG. Transforming and epidermal growth factors in degenerated intervertebral discs. J Bone Joint Surg Br. 1999 Nov;81(6):1058-63. doi: 10.1302/0301-620x.81b6.9321. PMID 10615986
- [Background] Wang SZ, Chang Q, Lu J, Wang C. Growth factors and platelet-rich plasma: promising biological strategies for early intervertebral disc degeneration. Int Orthop. 2015 May;39(5):927-34. doi: 10.1007/s00264-014-2664-8. Epub 2015 Feb 5. PMID 25653173
- [Background] Tolonen J, Gronblad M, Vanharanta H, Virri J, Guyer RD, Rytomaa T, Karaharju EO. Growth factor expression in degenerated intervertebral disc tissue. An immunohistochemical analysis of transforming growth factor beta, fibroblast growth factor and platelet-derived growth factor. Eur Spine J. 2006 May;15(5):588-96. doi: 10.1007/s00586-005-0930-6. Epub 2005 Jun 25. PMID 15980999
- [Background] Fujita N, Imai J, Suzuki T, Yamada M, Ninomiya K, Miyamoto K, Iwasaki R, Morioka H, Matsumoto M, Chiba K, Watanabe S, Suda T, Toyama Y, Miyamoto T. Vascular endothelial growth factor-A is a survival factor for nucleus pulposus cells in the intervertebral disc. Biochem Biophys Res Commun. 2008 Jul 25;372(2):367-72. doi: 10.1016/j.bbrc.2008.05.044. Epub 2008 May 19. PMID 18492486
- [Background] Civinini R, Macera A, Nistri L, Redl B, Innocenti M. The use of autologous blood-derived growth factors in bone regeneration. Clin Cases Miner Bone Metab. 2011 Jan;8(1):25-31. PMID 22461800
- [Background] Anitua E, Andia I, Ardanza B, Nurden P, Nurden AT. Autologous platelets as a source of proteins for healing and tissue regeneration. Thromb Haemost. 2004 Jan;91(1):4-15. doi: 10.1160/TH03-07-0440. PMID 14691563
- [Background] Hoogendoorn RJ, Lu ZF, Kroeze RJ, Bank RA, Wuisman PI, Helder MN. Adipose stem cells for intervertebral disc regeneration: current status and concepts for the future. J Cell Mol Med. 2008 Dec;12(6A):2205-16. doi: 10.1111/j.1582-4934.2008.00291.x. Epub 2008 Feb 24. PMID 18298653
- [Background] Masuda K, Oegema TR Jr, An HS. Growth factors and treatment of intervertebral disc degeneration. Spine (Phila Pa 1976). 2004 Dec 1;29(23):2757-69. doi: 10.1097/01.brs.0000146048.14946.af. PMID 15564925
- [Background] Pirvu TN, Schroeder JE, Peroglio M, Verrier S, Kaplan L, Richards RG, Alini M, Grad S. Platelet-rich plasma induces annulus fibrosus cell proliferation and matrix production. Eur Spine J. 2014 Apr;23(4):745-53. doi: 10.1007/s00586-014-3198-x. Epub 2014 Jan 28. PMID 24469887
- [Background] Tuakli-Wosornu YA, Terry A, Boachie-Adjei K, Harrison JR, Gribbin CK, LaSalle EE, Nguyen JT, Solomon JL, Lutz GE. Lumbar Intradiskal Platelet-Rich Plasma (PRP) Injections: A Prospective, Double-Blind, Randomized Controlled Study. PM R. 2016 Jan;8(1):1-10; quiz 10. doi: 10.1016/j.pmrj.2015.08.010. Epub 2015 Aug 24. PMID 26314234
- [Background] Pettine KA, Murphy MB, Suzuki RK, Sand TT. Percutaneous injection of autologous bone marrow concentrate cells significantly reduces lumbar discogenic pain through 12 months. Stem Cells. 2015 Jan;33(1):146-56. doi: 10.1002/stem.1845. PMID 25187512
- [Background] Pauza KJ, Howell S, Dreyfuss P, Peloza JH, Dawson K, Bogduk N. A randomized, placebo-controlled trial of intradiscal electrothermal therapy for the treatment of discogenic low back pain. Spine J. 2004 Jan-Feb;4(1):27-35. doi: 10.1016/j.spinee.2003.07.001. PMID 14749191
- [Background] Boswell MV, Trescot AM, Datta S, Schultz DM, Hansen HC, Abdi S, Sehgal N, Shah RV, Singh V, Benyamin RM, Patel VB, Buenaventura RM, Colson JD, Cordner HJ, Epter RS, Jasper JF, Dunbar EE, Atluri SL, Bowman RC, Deer TR, Swicegood JR, Staats PS, Smith HS, Burton AW, Kloth DS, Giordano J, Manchikanti L; American Society of Interventional Pain Physicians. Interventional techniques: evidence-based practice guidelines in the management of chronic spinal pain. Pain Physician. 2007 Jan;10(1):7-111. PMID 17256025
- [Background] Slosar PJ, Reynolds JB, Schofferman J, Goldthwaite N, White AH, Keaney D. Patient satisfaction after circumferential lumbar fusion. Spine (Phila Pa 1976). 2000 Mar 15;25(6):722-6. doi: 10.1097/00007632-200003150-00012. PMID 10752105
- [Background] Hedlund R, Johansson C, Hagg O, Fritzell P, Tullberg T; Swedish Lumbar Spine Study Group. The long-term outcome of lumbar fusion in the Swedish lumbar spine study. Spine J. 2016 May;16(5):579-87. doi: 10.1016/j.spinee.2015.08.065. Epub 2015 Sep 9. PMID 26363250
- [Background] Lee JJ, Lee MK, Kim JE, Kim HZ, Park SH, Tae JH, Choi SS. Pain relief scale is more highly correlated with numerical rating scale than with visual analogue scale in chronic pain patients. Pain Physician. 2015 Mar-Apr;18(2):E195-200. PMID 25794219
- [Background] Frost H, Lamb SE, Stewart-Brown S. Responsiveness of a patient specific outcome measure compared with the Oswestry Disability Index v2.1 and Roland and Morris Disability Questionnaire for patients with subacute and chronic low back pain. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2450-7; discussion 2458. doi: 10.1097/BRS.0b013e31818916fd. PMID 18824951